CLINICAL TRIAL: NCT03806426
Title: Randomised, Double-blind, Placebo-controlled Study of the Efficacy, Safety and Tolerability of EPA-FFA Gastro-resistant Capsules, in Patients With Familial Adenomatous Polyposis (FAP)
Brief Title: Effect of EPA-FFA on Polypectomy in Familial Adenomatous Polyposis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: S.L.A. Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPA-POL-04
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Eicosapentaenoic Acid; EPA; EPA 99%; Fatty Acid; omega-3; polyp; Familial Adenomatous Polyposis; FAP; IRA (Ileo-rectal anastomosis); PUFA (polyunsaturated fatty acid); Endoscopy
MeSH Terms: conditions — Adenomatous Polyposis Coli; Polyps | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group A (Experimental): Eicosapentaenoic acid free fatty acid (EPA-FFA) 500mg
  Interventions: Drug: Eicosapentaenoic acid free fatty acid (EPA-FFA)
- Treatment Group B (Placebo Comparator): Placebo 500mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eicosapentaenoic acid free fatty acid (EPA-FFA) — 500mg capsule, two 500mg capsules to be taken twice daily for 24 months
  Other Names: ALFA
  Arms: Treatment Group A
Drug: Placebo — 500mg capsule, two 500mg capsules to be taken twice daily for 24 months
  Arms: Treatment Group B

SUMMARY:
2 Year randomised, double-blind, placebo-controlled, parallel group study to determine the safety and efficacy of EPA-FFA gastro resistant capsules in FAP.

DETAILED DESCRIPTION:
The purpose of this Phase III study is to determine whether Eicosapentaenoic acid-free fatty acid is a safe and well tolerated treatment in reducing the number of polypectomies FAP patients with an APC gene mutation have over a 2 year treatment period and to assess the effect that this has on clinical disease progression. Planned Sample Size This study will enrol 204 subjects (102 subjects per treatment group). Primary Objective is to determine the efficacy of EPA-FFA gastro-resistant capsules in patients with FAP in reducing polypectomy.

Secondary objectives is to evaluate the clinical disease progression and the long-term safety and tolerability of EPA-FFA.

ELIGIBILITY:
Inclusion Criteria

1. Must give written informed consent.
2. Male or female subjects, 18 to 65 years of age.
3. Known diagnosis of FAP defined as those with a pathogenic APC mutation
4. Patients have had a previous colectomy with an ileo-rectal anastomosis or an ileal pouch- anal anastomosis with a rectal remnant of ≥ 2cm.
5. Classified stage 1-3 on InSiGHT Polyposis Staging System (IPSS).
6. Subjects must show a willingness to abstain from regular use of non-steroidal anti-inflammatory medication for the trial. A cardio protective dose of aspirin (75mg-100mg) will be permitted.

Exclusion Criteria:

1. Subjects with ileo-rectal anastomosis who have ≥ 20 polyps which are of >5mm that are not amendable to removal in the rectum.
2. Subjects unwilling to have regular sigmoidoscopy examination.
3. Subjects who are due to undergo gastro-intestinal surgery related to FAP.
4. History of invasive carcinoma in the past 3 years.
5. History of pelvic radiation.
6. Known allergic reaction or intolerant to fish or fish oils.
7. Known allergic reaction to excipients of IMP and placebo.
8. Subjects who are pregnant or breast-feeding at screening.
9. Subjects taking aspirin, other than a low (75mg-100mg) cardioprotective dose on a regular basis, or other nonsteroidal anti-inflammatory drugs (NSAIDs) on a regular basis. Regular use of other NSAIDS is defined in this protocol as use greater than 14-day treatment period, and one treatment per six months for the duration of the study.
10. Subjects taking NSAIDs regularly in the 3 months prior to entry (other than low dose aspirin).
11. Subjects taking NSAID, 5-aminosalicylic acid (5-ASA or mesalamine).
12. Subjects who are taking other fish-oil supplements (e.g. cod liver oil) who are unwilling to stop them for the duration of the study. Subjects previously taking fish oil must have a washout period of 2 months prior to study enrolment.
13. Subjects who are taking warfarin or other anticoagulants.
14. Experimental agents must have been discontinued at least 8 weeks prior to screening or for a period equivalent to 5 half-lives of the agent (whichever is longer).
15. Subjects suffering from known disorders of clotting and blood coagulation.
16. Subjects who have significant abnormalities on their screening blood tests.
17. Subjects with gastrointestinal malabsorptive disease.
18. Subjects with uncontrolled hypercholesterolaemia.
19. Subjects who are deemed mentally incompetent or have a history of anorexia nervosa or bulimia.
20. Subjects who will be unavailable for the duration of the trial, deemed unable to comply with the requirements of the study protocol, likely to be noncompliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason.
21. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless surgically sterile, must use effective contraception (either combined oestrogen and progestogen containing hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD], intrauterine hormone-releasing system [IUS], vasectomised partner, sexual abstinence (only considered an acceptable method of contraception when it is in line with the subjects' usual and preferred lifestyle), combination of male condom with either cap, diaphragm or sponge with spermicide [double barrier methods]), and willing and able to continue contraception for 1 month after the last administration of IMP.
22. Women using oral contraception must have started using it at least 2 months prior to screening. Women are not considered to be of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels that have been confirmed to be in the "postmenopausal range". Or have had a surgical bilateral oophorectomy (with or without hysterectomy) or bilateral tubal ligation at least six weeks before the screening visit. In case of oophorectomy alone, the reproductive status of the woman should have been confirmed by follow up hormone level assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Total Number of Polypectomies (polyps > 5mm in the rectum) conducted during the 24 months study period | 24 months
  Proctectomy is indicated when polyp burden is frequently high in the remaining rectum, if large highly dysplastic polyps occur, or if frank malignancy develops. Proctocolectomy also significantly reduces the cancer risk with the removal of the colon and rectum.

SECONDARY OUTCOMES:
Change in Polyp number at 24 months assessed by blinded review of video records | 24 months
  Subsequent proctectomy is indicated when polyp burden is frequently high in the remaining rectum, if large highly dysplastic polyps occur, or if frank malignancy develops. Proctocolectomy also significantly reduces the cancer risk with the removal of the colon and rectum.
Change in score on the InSIGHT Polyposis Staging System (IPSS) at 24 months | 24 months
  Classified stage on InSiGHT Polyposis Staging System (IPSS). The subjects FAP will be classified in accordance with the IPSS.
  The IPSS classification will be verified by the Polyp Video Scoring committee

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ricciardiello, MD, Principal Investigator — Associate Professor of Gastroenterology, University of Bologna
Locations (1):
- University of Bologna and St.Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No